CLINICAL TRIAL: NCT04229771
Title: Does Administration of Proparacaine Hydrochloride 0.5% Ophthalmic Solution Prior to Canalicular Probing and Irrigation Decrease Patient Discomfort
Brief Title: Does Topical Ophthalmic Anesthetic Prior to Probing and Irrigation Decrease Pain?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Dianne Schlachter MD, Principal Investigator, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-216
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Epiphora; Dacryostenosis; Dacryocystitis
Keywords: Nasolacrimal duct obstruction; Probe and irrigation
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Dacryocystitis; Lacrimal Duct Obstruction | interventions — proxymetacaine; Hanks Balanced Salt Solution

STUDY DESIGN:
Intervention Model Description: A double-blinded, randomized, controlled clinical trial with one eye of each participant receiving the experimental treatment and one eye acting as control, receiving placebo
Who Masked: Participant, Care Provider
Masking Description: Randomization will be performed by the primary investigator who will have no participant interaction during the performance of the procedure and obtainment of the survey responses. A random number generator will be used to obtain either an even or odd number. Odd numbers mean the left eye receives Proparacaine hydrochloride 0.5% ophthalmic solution, even numbers mean the right eye does. The chief investigator will instruct clinic personnel as to which syringe should be labeled "L" or "R" depending on randomization results.Two identical 1 ml syringes will be prepared. One syringe containing control BSS, and the other containing Proparacaine hydrochloride 0.5% ophthalmic solution. Each syringe will be labeled by clinical assistants with either left (L) or right (R) as randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Participants who received proparacaine hydrochloride solution in left eye and placebo in right eye (Experimental): Participants receiving a drop of Proparacaine Hydrocholoride 0.5% ophthalmic solution in left eye and a drop of basic salt solution (BSS, placebo) in the right eye prior to probing and irrigation.
  Interventions: Drug: Proparacaine Hydrochloride ophthalmic solution, USP 0.5%; Drug: Balanced salt solution
- Participants who received proparacaine hydrochloride solution in right eye and placebo in left eye (Experimental): Participants receiving a drop of Proparacaine Hydrocholoride 0.5% ophthalmic solution in right eye and a drop of basic salt solution (BSS, placebo) in the left prior to probing and irrigation.
  Interventions: Drug: Proparacaine Hydrochloride ophthalmic solution, USP 0.5%; Drug: Balanced salt solution

INTERVENTIONS:
Drug: Proparacaine Hydrochloride ophthalmic solution, USP 0.5% — One drop instilled in one eye, randomly chosen, as topical anesthetic
  Other Names: Alcaine
Drug: Balanced salt solution — One drop instilled in one eye, randomly chosen, as control placebo
  Other Names: BSS

SUMMARY:
Purpose: It is unknown whether instillation of a drop of anesthetic ophthalmic solution into the eye such as proparacaine hydrochloride 0.5% prior to probing and irrigation of the tear duct (lacrimal drainage) system improves participant comfort during the procedure. To date, there have been no formal studies evaluating the possible benefit of this pretreatment.

Methods: Participants 18 years and older who present to the William Beaumont Hospital - Royal Oak, Michigan outpatient ophthalmology clinic with a chief complaint of epiphora (excessive tearing) who necessitate bilateral lower lid probing and irrigation of the lacrimal drainage system will be enrolled in the study. One eye will be randomized to receive a drop of the anesthetic Proparacaine hydrochloride 0.5% and the other eye will receive a control drop of Balanced Salt Solution (BSS). Probing and irrigation will then be performed in the usual fashion. The participant will then be questioned via survey on a pain scale of 1-5 as to the amount of subjective pain experienced on each side during the procedure.

Expected Results: Investigators expect participants will experience statistically significantly less pain in eyes that have received a drop of Proparacaine hydrochloride 0.5% prior to performance of probing and irrigation compared to the eyes which have received the control drop.

DETAILED DESCRIPTION:
Rationale: It is common for male and female adults of all races with a chief complaint of epiphora (excessive tearing) to express discomfort either verbally or through body language while undergoing tear duct (canalicular) probing and irrigation even when no pathology is detected. Use of a topical anesthetic during canalicular probing and irrigation is seen in children but has yet to be formally investigated in adults to date. The goal of this study is to identify whether or not instillation of a drop of Proparacaine hydrochloride 0.5% ophthalmic solution into a participant's eye prior to performance of probing and irrigation will improve participant comfort during the procedure and is therefore recommended.

Hypothesis: Administration of a drop of Proparacaine hydrochloride 0.5% ophthalmic solution into the eye prior to probing and irrigation of the lower lid canalicular system will decrease discomfort as compared to a control drop of BSS ophthalmic solution into the opposite eye prior to the same procedure.

Null hypothesis: Administration of a drop of Proparacaine hydrochloride 0.5% ophthalmic solution does not have an effect on discomfort during canalicular probing and irrigation.

Medication: Proparacaine hydrochloride ophthalmic solution, United States Pharmacopeia (USP) 0.5% is a local anesthetic drug intended for topical ophthalmic use. Proparacaine Hydrochloride ophthalmic solution is a fast-acting anesthetic lasting 10-20 minutes. Proparacaine hydrochloride ophthalmic solution, USP 0.5% is FDA approved for this indication.

Probing and irrigation: A common in-office ophthalmic procedure performed with a small gauge, blunt tube on a syringe filled with BSS. The cannula is placed into the canaliculus (tear duct) of one eyelid, and the BSS is used to irrigate the lacrimal system. This procedure identifies whether or not obstruction of the lacrimal system is present. A participant with an open (patent) system will taste the salty BSS solution in the nose. A participant with a nasolacrimal duct obstruction (NLDO) or a more proximal canalicular obstruction will have reflux of the irrigant out of the opposite lid (on the same side) canaliculus, the probed canaliculus, or both and will usually not detect any irrigant within the nasopharynx.

Definitions:

Nasolacrimal drainage system: The physiologic apparatus which drains tears from the surface of the eye into the nose (i.e. the tear drain). It consists of (from eye to nose) the punctum (opening of the tube), the canaliculus (a thin tube within the eyelid), the lacrimal sac (a sac that hold the tears that lies within the bone of the nose) and finally the nasolacrimal duct (a duct that connects the lacrimal sac (-lacrimal) into the nose (naso-). A blockage anywhere along this pathway can cause epiphora.

Epiphora: The pathological process of tears overflowing from the ocular surface and rolling down the face. Commonly caused by obstructions of the lacrimal drainage system. Can cause significant irritation and loss of vision.

ELIGIBILITY:
Inclusion Criteria:

* Participants of any sex aged 18 years or older
* Signs and symptoms of epiphora which necessitate performance of a diagnostic probing and irrigation of the bilateral lower eyelid lacrimal drainage system at Beaumont Royal Oak or any of the listed physician offices who present with a chief complaint of epiphora from either eye

Exclusion Criteria:

* A known allergy to topical proparacaine hydrochloride
* Known pre-existing scarring, surgery, radiation to the nasolacrimal system
* Presence of blockage and or reflux on probing and irrigation of either side
* Cognitive Impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dianne M Schlachter, MD, Principal Investigator — Corewell Health East
Locations (1):
- Dianne Schlachter, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data to be shared

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Who Received Proparacaine Hydrochloride Solution in Left Eye and Placebo in Right Eye: Participants will have received a drop of Proparacaine Hydrocholoride 0.5% ophthalmic solution in left eye and a drop of basic salt solution (BSS, placebo) in the right eye prior to probing and irrigation.
  Proparacaine Hydrochloride ophthalmic solution, United States Pharmacopeia (USP) 0.5%: One drop instilled in left eye, as topical anesthetic
  Balanced salt solution: One drop instilled in right eye, as control placebo
- Participants Who Received Proparacaine Hydrochloride Solution in Right Eye and Placebo in Left Eye: Participants will have received a drop of Proparacaine Hydrocholoride 0.5% ophthalmic solution in right eye and a drop of basic salt solution (BSS, placebo) in the left prior to probing and irrigation.
  Proparacaine Hydrochloride ophthalmic solution, United States Pharmacopeia (USP) 0.5%: One drop instilled in right eye, as topical anesthetic
  Balanced salt solution: One drop instilled in left eye, as control placebo
Period: Overall Study
Arm/Group | Participants Who Received Proparacaine Hydrochloride Solution in Left Eye and Placebo in Right Eye | Participants Who Received Proparacaine Hydrochloride Solution in Right Eye and Placebo in Left Eye
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants randomized to the group "Participants who received proparacaine hydrochoride solution in the right eye and placebo in the left eye."
Units Other Than Participants: eyes
Groups:
- Participants Who Received Proparacaine Hydrochloride Solution in Left Eye and Placebo in Right Eye: Participants will have received a drop of Proparacaine Hydrocholoride 0.5% ophthalmic solution in left eye and a drop of balanced salt solution (BSS, placebo) in the right eye prior to probing and irrigation.
  Proparacaine Hydrochloride ophthalmic solution, USP 0.5%: One drop instilled in left eye, as topical anesthetic
  Balanced salt solution: One drop instilled in right eye, as control placebo
- Participants Who Received Proparacaine Hydrochloride Solution in Right Eye and Placebo in Left Eye: Participants will have received a drop of Proparacaine Hydrocholoride 0.5% ophthalmic solution in right eye and a drop of balanced salt solution (BSS, placebo) in the left prior to probing and irrigation.
  Proparacaine Hydrochloride ophthalmic solution, USP 0.5%: One drop instilled in right eye, as topical anesthetic
  Balanced salt solution: One drop instilled in left eye as control placebo
- Total: Total of all reporting groups
Arm/Group | Participants Who Received Proparacaine Hydrochloride Solution in Left Eye and Placebo in Right Eye | Participants Who Received Proparacaine Hydrochloride Solution in Right Eye and Placebo in Left Eye | Total
Number analyzed (Participants) | 2 | 0 | 2
Number analyzed (eyes) | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (7.7) |  | 69.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 1 |  | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Who Report of Less Discomfort in the Eye That Received the Proparacaine Hydrochloride Anesthetic During Probing
Description: Participants completed a survey which asked which procedure was more uncomfortable (left or right). Assignment to receive proparacaine hydrochloride was compared to survey results. When the participant reported less discomfort in the eye that received the proparacaine hydrochloride medication, this is is reported as concordance between reduction of pain/discomfort and anesthetic use.
Time Frame: 1 minute
Population: No participants were randomized to arm "Participants who received proparacaine hydrochloride in right eye and placebo in left eye."
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Received Proparacaine Hydrochloride Solution in Left Eye and Placebo in Right Eye: Participants will have received a drop of Proparacaine Hydrocholoride 0.5% ophthalmic solution in left eye and a drop of balanced salt solution (BSS, placebo) in the right eye prior to probing and irrigation.
  Proparacaine Hydrochloride ophthalmic solution, USP 0.5%: One drop instilled in left eye, as topical anesthetic
  Balanced salt solution: One drop instilled in right eye as control placebo
- Participants Who Received Proparacaine Hydrochloride Solution in Right Eye and Placebo in Left Eye: Participants will have received a drop of Proparacaine Hydrocholoride 0.5% ophthalmic solution in right eye and a drop of basic salt solution (BSS, placebo) in the left prior to probing and irrigation.
  Proparacaine Hydrochloride ophthalmic solution, USP 0.5%: One drop instilled in right eye, as topical anesthetic
  Balanced salt solution: One drop instilled in one eye, randomly chosen, as control placebo
Arm/Group | Participants Who Received Proparacaine Hydrochloride Solution in Left Eye and Placebo in Right Eye | Participants Who Received Proparacaine Hydrochloride Solution in Right Eye and Placebo in Left Eye
Number analyzed (Participants) | 2 | 0
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: Number at risk for Serious Adverse Events, All-Cause Mortality and Other (Not including Serious) Adverse Events is zero for the group "Participants who Received Proparacaine Hydrochloride Solution in Right Eye" because no participants were randomized to this arm.
Groups:
- Participants Who Received Proparacaine Hydrochloride Solution in Left Eye and Placebo in Left Eye: Participants will have received a drop of Proparacaine Hydrocholoride 0.5% ophthalmic solution in left eye and a drop of basic salt solution (BSS, placebo) in the right eye prior to probing and irrigation.
  Proparacaine Hydrochloride ophthalmic solution, USP 0.5%: One drop instilled in left eye, as topical anesthetic
  Balanced salt solution: One drop instilled in right eye, as control placebo
- Participants Who Received Proparacaine Hydrochloride Solution in Right Eye and Placebo in Left Eye: Participants will have received a drop of Proparacaine Hydrocholoride 0.5% ophthalmic solution in right eye and a drop of basic salt solution (BSS, placebo) in the left prior to probing and irrigation.
  Proparacaine Hydrochloride ophthalmic solution, USP 0.5%: One drop instilled right eye, as topical anesthetic
  Balanced salt solution: One drop instilled in left eye, as control placebo
Arm/Group | Participants Who Received Proparacaine Hydrochloride Solution in Left Eye and Placebo in Left Eye | Participants Who Received Proparacaine Hydrochloride Solution in Right Eye and Placebo in Left Eye
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT04229771/Prot_SAP_001.pdf